CLINICAL TRIAL: NCT06989190
Title: The MIND Study - Microangiopathy IN Diabetes
Status: Recruiting | Type: Observational
Sponsor: HJN Sverige AB/Neko Health (Industry)
Responsible Party: Sponsor
Other Study IDs: CIV-23-02-042193
Record Dates: First submitted 2025-05-08; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A total of 30 ml och blood/plasma is saved for each study subject for later research analyses. Research blood samples are saved as whole blood or centrifuged directly at the Danderyd Department of Clinical Sciences laboratory, and is saved in smaller aliquotes (á 205 or 500 uL) which are marked with the study subject's pseudonymised participant ID/code number. Samples are kept in a -80 °C freezer at Danderyd Hospital under Stockholms Medicinska Biobank (SMD, reg nr 914) with Stockholm Municipality as the responsible party.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- diabetes_severe_cohort: Patients with severe type 1 diabetes (microangiopathy / diabetic feet), with complications. Severe angiopathy defined as proliferative retinopathy, macroalbuminuria, and kidney failure with at least CKD-class 3B and severe neuropathy with or without foot ulcers.
- diabetes_moderate_cohort: Patients with type 1 diabetes and moderate microangiopathy. moderate non-proliferative retinopathy or proliferative retinopathy, macroalbuminuria or kidney failure (defined as estimated glomerular filtration rate <60 mL/min/1.73 m2 body surface) up to CKD-class 3A, and manifest neuropathy, (group c).
- diabetes_mild_cohort: Patient with mild microangiopathy, mild-moderate non-proliferative retinopathy and/or microalbuminuria and/or early signs of neuropathy (group b).
- diabetes_none_cohort: Patient with no microangiopathy, except for simplex or background retinopathy, which is in an early and reversible state (group a).
- healthy_cohort: Age- and sex- matched healthy controls, with no known increased risk of cardiovascular disease.

SUMMARY:
This clinical investigation will evaluate two contactless optical devices based on spatial frequency domain and laser speckle technology for quantification of the skin micro-circulation in patients with diabetes mellitus type 1.

DETAILED DESCRIPTION:
This clinical feasibility study aims to evaluate the potential of contactless and non-invasive technologies for measurement of skin microcirculatory properties and their regulatory function in healthy individuals and patients with diabetes type 1. The clinical investigation incorporates two investigational devices:

* Neko Health TCI P4: a contactless optical device based on SFDI technology, to be used for quantification of the skin microcirculation via molecular composition, such as haemoglobin / blood volume and oxygen concentrations.
* Perimed Multiflow: a contactless optical device based on laser speckle technology, to be used for quantification of the skin micro-circulation via speed resolved perfusion based on movement of the red blood cells.

These technologies are promising tools for diagnostic support of pathology in the microcirculation, such as diabetic microangiopathy. Since they are imaging technologies, collecting data over a two-dimensional surface of the skin; they may be more robust than single-point measurements as well as allowing for quantification of differences and distribution over different skin sections.

The two investigational devices are good complements, as the TCI P4 can quantify composition (concentration of molecules) and the MultiFlow can quantify flow properties (perfusion), this way one gets a good foundation to study the key properties of the micro-circulation: blood volume, oxygenation and hemodynamics.

The state of the art concerning diabetic complications and PAD (Peripheral Arterial Disease) in clinical practice is currently not proactive, but rather aimed towards reactive treatment, management, and monitoring during the later phase of tissue damage and microvascular impairment. The aim with the investigation is to find indication of disease / pathology at an early stage, by evaluation of parameters / physiological changes before manifestation of clinical complications. The state-of-the-art guidelines on diagnosis, prognosis, and management of PAD in patients with foot ulcers and diabetes are well described in the 2023 WGDF Guidelines on the Prevention and Management of Diabetes-related Foot Disease. These guidelines are based on pressure-based measurements, ABI (Ankle Brachial Index), TBI (Toe Brachial Index) and tcpO2. The pathophysiological features of PAD and diabetes foot ulcers is primarily due to altered blood perfusion and tissue oxygenation whereas the investigational device is assessing the micro-circulation (smaller vessels). However, since the micro-circulation is connected downstream to the larger vessels (macro-circulation) its perfusion will be affected by both macro- and micro-circulatory factors. Therefore, the investigational device may enable finding early indications of pathology regardless of if the issue starts in the macro- or micro-circulation. Furthermore, micro-circulatory changes correlated to PAD and diabetes in skin tissue has been proven in published research, for skin in feet [1], as well as skin in the forearm [2], [3].

The hypotheses will be analysed by correlation analysis (simple regression coefficients) between physiological response and the measured parameters, along with other analytical methods suitable for understanding these correlations. Interpretation of the observed physiological response will be based on theoretical background as well as results from the comparator devices. Data of patients with diabetes type 1 and different severities of clinical microangiopathy will be compared to healthy controls, in order to see if responses are altered by diabetes microangiopathy and if they can be isolated from normal variation in the control group.

Furthermore, the hypothesis is also that different body sites are affected differently and at different stages of pathology, due to the local properties and environment of the different sites. The relation in properties between the sites may also be altered by diabetes microangiopathy. For example, peripheral body sites are usually seen to be affected first by pathology. The following body sites will be investigated:

* Volar side of forearm
* Palm of hand
* Dorsal and plantar side of feet

The main outcomes are listed below, however all generated datatypes of each examination will be analysed for any correlations between them and the status of the patient, to ensure that important correlations and learnings are not missed, even if the specific correlation was not expected.

ELIGIBILITY:
Phase 1: Severe Diabetic Complications (50 patients)

Inclusion Criteria:

* Severe type 1 diabetes (microangiopathy / diabetic feet), severe angiopathy defined as proliferative retinopathy, macroalbuminuria, and kidney failure with at least CKD-class 3B and severe neuropathy with or without foot ulcers.
* Age range: primarily 18-45 years, if not sufficient number of subjects can be found, then 18-60 years span is considered

Phase 2: Scale of severity. In phase 2, patients are included with a broad range of severity levels. Patients with diabetes type 1 will be included.

Inclusion criteria:

* Age range: 18-45 years (younger patients are targeted for focus on microvascular complications, rather than age-related cardiovascular disease)
* Patient with no microangiopathy, except for simplex or background retinopathy, which is in an early and reversible state (group a), 100 patients.
* Patient with mild microangiopathy, mild-moderate non-proliferative retinopathy and/or microalbuminuria and/or early signs of neuropathy (group b), 100 patients.
* Patient with moderate microangiopathy. moderate non-proliferative retinopathy or proliferative retinopathy, macroalbuminuria or kidney failure (defined as estimated glomerular filtration rate <60 mL/min/1.73 m2 body surface) up to CKD-class 3A, and manifest neuropathy, (group c), 50 patients.

Healthy controls:

- Healthy control matched to the type 1 diabetes patients in age and gender, with no known risk of increased cardiovascular disease.

Exclusion Criteria:

* Patients unable to understand patient information due to cognitive impairment
* Patients unable to understand patient information due to language barriers
* Ongoing acute infection or inflammatory condition
* Pregnant or breastfeeding women
* Patients with damaged and/or scarred tissue in the areas of interest for the investigational or comparator devices

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with type 1 diabetes will be recruited from the diabetes clinic at Danderyd Hospital, which currently follows around 1800 patients with type 1 diabetes. All patients matching the inclusion criteria will be asked to participate in the study by a doctor or nurse at their routine visit to the clinic. Responsible doctor or research nurse will also screen for suitable patients registered at the clinic, and call the patients that meet inclusion criteria to see if they would like to participate in the study after a short description of the study's purpose and setup.
  Recruitment of the control group will occur through digital advertisement, e.g. on the Karolinska Institute website.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between investigational device-derived energy in endothelial band and endothelial pathology | Same day as enrolment.
  Correlation between SFDI- and laser speckle-derived endothelial energy band (perfusion, oxygenation) and blood marker indication of endothelial cell /glycocalyx deterioration and/or endothelial cell response from iontophoresis provocation.
Correlation between investigational device-derived energy in the myogenic band in the case of hypertension and myogenic related pathology | Same day as enrolment.
  Association between SFDI- and laser speckle-derived myogenic energy band and presence of hypertension, and/or indication of reduced smooth muscle cell response from iontophoresis provocation.
Correlation between investigational device-derived energy in the neurogenic band and indication of neuropathy | Same day as enrolment.
  Correlation between SFDI- and laser speckle-derived neurogenic energy band and indication/diagnosis of neuropathy, based on clinical assessment or electronic health records.
Correlation between investigational device-derived brachial post-occlusive hyperemia (PORH) peak oxygenation and degree of neuropathic angiopathy | Same day as enrolment.
  Correlation of investigational device-derived peak oxygen saturation amplitude from brachial PORH test against degree of microangiopathy/ microvascular complications.
Difference in response (perfusion) to mild local heat provocation between diabetes type 1 and healthy controls | Same day as enrolment.
  Difference in IMD-derived variables of perfusion between healthy controls and patients with diabetes type 1 during mild local heat provocation (~30ᵒC).
Difference in response (oxygenation) to mild local heat provocation between diabetes type 1 and healthy controls | Same day as enrolment.
  Difference in IMD-derived variables of oxygenation between healthy controls and patients with diabetes type 1 during mild local heat provocation (~30ᵒC).
Difference in response (hemoglobin concentration) to mild local heat provocation between diabetes type 1 and healthy controls | Same day as enrolment.
  Difference in IMD-derived variables of hemoglobin concentration between healthy controls and patients with diabetes type 1 during mild local heat provocation (~30ᵒC).
Difference in response (perfusion) to increased local heat provocation between diabetes type 1 and healthy controls | Same day as enrolment.
  Difference in IMD-derived variables of perfusion between healthy controls and patients with diabetes type 1 during increased local heat provocation (~35ᵒC).
Difference in response (oxygenation) to increased local heat provocation between diabetes type 1 and healthy controls | Same day as enrolment.
  Difference in IMD-derived variables of oxygenation between healthy controls and patients with diabetes type 1 during increased local heat provocation (~35ᵒC).
Difference in response (hemoglobin concentration) to increased local heat provocation between diabetes type 1 and healthy controls | Same day as enrolment.
  Difference in IMD-derived variables of hemoglobin concentration between healthy controls and patients with diabetes type 1 during increased local heat provocation (~35ᵒC).
Difference in response (perfusion) to high local heat provocation between diabetes type 1 and healthy controls | Same day as enrolment.
  Difference in IMD-derived variables of perfusion between healthy controls and patients with diabetes type 1 during high local heat provocation (~40-44ᵒC).
Difference in response (oxygenation) to high local heat provocation between diabetes type 1 and healthy controls | Same day as enrolment.
  Difference in IMD-derived variables of oxygenation between healthy controls and patients with diabetes type 1 during high local heat provocation (~40-44ᵒC).

SECONDARY OUTCOMES:
Assessment of distribution of oxygenation in foot soles of patients with diabetic feet compared to healthy controls | Same day as enrolment.
  Comparison of the distribution oxygenation on the foot sole in diabetic feet of risk level 2-4 (levels as set by national guidelines) and feet of healthy controls with no evidence of cardiovascular disease.
Assessment of distribution of perfusion in foot soles of patients with diabetic feet compared to healthy controls | Same day as enrolment.
  Comparison of the distribution of perfusion on the foot sole in diabetic feet of risk level 2-4 (levels as set by national guidelines) and feet of healthy controls with no evidence of cardiovascular disease.
Assessment of if the addition of thermal provocation can increase contrasts between diabetic feet and feet of healthy controls | Same day as enrolment.
  Comparison of the distribution during response to heat provocation in diabetic feet compared to feet of healthy controls to assess contribution to differences between groups.
Assessment of if the addition of investigational device-derived water concentration data can increase contrasts between diabetic feet and feet of healthy controls | Same day as enrolment.
  Comparison of the distribution of other variables such as SFDI-derived water concentration in diabetic feet compared to feet of healthy controls to assess contribution to differences between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Tehrani, MD, PhD, Principal Investigator — Danderyd Hospital, Department of Internal Medicine, Stockholm, Sweden
Locations (1):
- VO Medicinska Specialiteter, Danderyd Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Jonasson H, Bergstrand S, Fredriksson I, Larsson M, Ostgren CJ, Stromberg T. Post-ischemic skin peak oxygen saturation is associated with cardiovascular risk factors: a Swedish cohort study. Microvasc Res. 2022 Mar;140:104284. doi: 10.1016/j.mvr.2021.104284. Epub 2021 Nov 23. PMID 34826433
- [Background] Murphy GA, Singh-Moon RP, Mazhar A, Cuccia DJ, Rowe VL, Armstrong DG. Quantifying dermal microcirculatory changes of neuropathic and neuroischemic diabetic foot ulcers using spatial frequency domain imaging: a shade of things to come? BMJ Open Diabetes Res Care. 2020 Nov;8(2):e001815. doi: 10.1136/bmjdrc-2020-001815. PMID 33219118